CLINICAL TRIAL: NCT05458388
Title: Different Endoscopic Gastric Cancer Risk Assessments for the Detection of Early Gastric Cancer
Brief Title: Different Endoscopic Gastric Cancer Risk Assessments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yanqing Li (Other)
Responsible Party: Sponsor-Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Organization: Shandong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2022-SDU-QILU-120
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Gastric Cancer Screening

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kimura-Takemoto classification (Active Comparator)
  Interventions: Procedure: Kimura-Takemoto classification
- EGGIM (Active Comparator)
  Interventions: Procedure: EGGIM

INTERVENTIONS:
Procedure: Kimura-Takemoto classification — All patients were given two risk scores, the order of which was randomly determined.
  Arms: Kimura-Takemoto classification
Procedure: EGGIM — All patients were given two risk scores, the order of which was randomly determined.
  Arms: EGGIM

SUMMARY:
The Kimura-Takamoto classification established in Japan can observe the extent of gastric atrophy in real-time under endoscopy, and diffuse atrophy also indicates an increased risk of gastric cancer. Recent studies have found that the evaluation of intestinal metaplasia score (EGGIM score) of various stomach parts by electronic staining can well identify OLGIM III\ IV patients. Although the Kimura-Takamoto classification and EGGIM score can evaluate the risk of gastric cancer in patients, only in cross-sectional studies, it is not clear the diagnostic value of risk assessment in population screening. Early gastric cancer has the characteristics of hidden lesions and a high rate of clinical missed diagnosis. Concentrating high-risk groups through risk scores is expected to guide endoscopic doctors to conduct a targeted careful examination. However, it is not clear whether Kimura-Takamoto classification and EGGIM score can improve the detection rate of early gastric cancer in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-80 years undergoing gastroscopy
* Patients intend to undergo ESD treatment

Exclusion Criteria:

* patients with severe cardiac, cerebral, pulmonary or renal dysfunction or psychiatric disorders who cannot participate in gastroscopy
* Patients with previous surgical procedures on the stomach
* patients with contraindications to biopsy
* Patients who refuse to sign the informed consent form.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-04 (Estimated)

PRIMARY OUTCOMES:
Early gastric cancer detection rate | 36 months
  The detection rate of early gastric cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China